CLINICAL TRIAL: NCT01855815
Title: HL-CA-1600, Hemolung RAS Registry. A Retrospective Registry Involving Voluntary Reporting of De-identified, Standard of Care Data Following the Commercial Use of the Hemolung Respiratory Assist System (RAS)
Brief Title: Hemolung RAS Registry Program
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Alung Technologies (Industry)
Responsible Party: Sponsor
Other Study IDs: HL-CA-1600
Record Dates: First submitted 2013-05-13; First posted 2013-05-17 (Estimated); Last update posted 2019-01-28 (Actual); Status verified 2019-01

CONDITIONS: Acute Hypercapnic Respiratory Failure
MeSH Terms: conditions — Respiratory Insufficiency

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of the Hemolung RAS Registry Program is to collect retrospective, de-identified, standard of care data following the commercial use of the Hemolung RAS.

DETAILED DESCRIPTION:
ALung's post-market Hemolung RAS Registry Program provides a continuum for measuring the Hemolung RAS effectiveness and safety in a real-world setting beyond the results reported in pre-market clinical feasibility studies. The Hemolung RAS Registry Program is part of ALung's 1) evaluation of clinical evidence throughout the life cycle of the product, 2) longer term residual risk assessment of the product, and 3) commitment to maintain quality systems and integrate continuous quality improvements in the product.

On a voluntary basis, participating physicians and institutional staff enter de-identified data online in the secure, password protected, regulatory-compliant Hemolung RAS Registry Portal in a retrospective manner following a patient's ICU discharge, status at 28 days post-Hemolung therapy, or death whichever is earlier. There is no requirement to collect and report data outside of standard of care. The program's methodology, data monitoring and statistical analysis plan is consistent with this type of initiative in a real-world setting.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Severe COPD or ARDS
Sampling Method: Non-Probability Sample
Enrollment: 99 (Estimated)
Dates: Start 2013-04; Primary Completion 2019-12 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
Number of days in the ICU | Patient data will only be reported for up to a maximum of 28 days from Hemolung therapy initiation.
Number of days on Hemolung therapy | Patient data will only be reported for up to a maximum of 28 days from Hemolung therapy initiation.
Incidents | Patient data will only be reported for up to a maximum of 28 days from Hemolung therapy initiation.
Outcome at 28 days | Patient data will only be reported for up to a maximum of 28 days from Hemolung therapy initiation.

SECONDARY OUTCOMES:
Patient mobility on Hemolung | Patient data will only be reported for up to a maximum of 28 days from Hemolung therapy initiation.
Blood product usage and hematologic effects on Hemolung | Patient data will only be reported for up to a maximum of 28 days from Hemolung therapy initiation.
Arterial blood gas changes on Hemolung | Patient data will only be reported for up to a maximum of 28 days from Hemolung therapy initiation.
Ventilatory mode and setting changes on Hemolung | Patient data will only be reported for up to a maximum of 28 days from Hemolung therapy initiation.
CO2 removal and blood flow performance | Patient data will only be reported for up to a maximum of 28 days from Hemolung therapy initiation.
Hemolung-assisted weaning | Patient data will only be reported for up to a maximum of 28 days from Hemolung therapy initiation.

CONTACTS AND LOCATIONS:
Overall Officials: Nausherwan Burki, MD, PhD, Study Director — ALung Technologies, Inc.